CLINICAL TRIAL: NCT05824520
Title: Coronary Computed Tomography-Derived Fraction Flow Reserve (FFR)-Guided Invasive Treatment Strategy (ITS) Versus Optimal Medical Therapy (OMT) Alone in Patient With Chronic Coronary Syndrome
Brief Title: Coronary CT-Derived FFR-Guided Strategy Versus Medical Therapy
Acronym: ACCURATE II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0318
Record Dates: First submitted 2023-03-06; First posted 2023-04-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Myocardial Ischaemia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-derived FFR guided-ITS group (Experimental): CT-derived FFR≤0.8; ITS plus OMT
  Interventions: Other: ITS plus OMT
- Medical therapy group (Active Comparator): CT-derived FFR≤0.8; OMT alone
  Interventions: Other: OMT

INTERVENTIONS:
Other: ITS plus OMT — Invasive treatment strategy plus optimal medical therapy
  Arms: CT-derived FFR guided-ITS group
Other: OMT — Optimal medical therapy alone
  Arms: Medical therapy group

SUMMARY:
The overall purpose of ACCURATE II trial is to compare the clinical outcomes of CT-derived FFR guided strategy versus medical therapy in patients with chronic coronary syndrome.

DETAILED DESCRIPTION:
ACCURATE II is a prospective, multicenter, randomized clinical trial comparing the clinical outcome and cost-effectiveness of the two management strategies. CT-FFR-guided invasive treatment strategy versus optimal medical therapy, in management of patients with chronic coronary syndrome. The study is powered to detect if the primary endpoint by the CT-FFR-guided strategy is superior to the medical therapy strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, with at least one vessel has CT-derived FFR≤0.80
* Patients with chronic coronary syndromes
* Signed written informed consent

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Contrast media (Patients with documented sensitivity to contrast media which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled)
* Prior percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Sinus arrhythmia, cardiogenic shock, or severe heart failure (NYHA≥III)
* Inability or unwillingness to undergo CT scan or coronary angiography
* Patients on hemodialysis or with severe hepatic or renal insufficiency
* Left main coronary artery stenosis ≥ 50%
* Target vessel total occlusion
* Pregnancy or intention to become pregnant during the course of the trial
* Patients with a life expectancy less than 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1066 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-10-20 (Estimated); Study Completion 2032-10-20 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 year
  A composite of all-cause death, myocardial infarction (MI) or ischemia-driven revascularization.

SECONDARY OUTCOMES:
Death | 1 year
  All-cause death and cardiac death.
MI | 1 year
  Target vessel related and non-target vessel related MI.
Revascularization | 1 year
  Ischemia driven, non-ischemia driven, target vessel and non-target vessel revascularization.
Stroke | 1 year
  Stroke (ischemic and hemorrhagic).
Cost-effectiveness analysis | 1 year
  Medical expenses of treatment and follow-up.
Quality of life assessed by Seattle Angina Questionnaire | 1 year
  Frequency of angina and the disease-specific quality of life, as assessed by Seattle Angina Questionnaire.
MACE | 1 month, 2 years, 3 years, 5 years
  A composite of all-cause death, myocardial infarction (MI) or ischemia-driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No